CLINICAL TRIAL: NCT00825279
Title: Comparison Among a Paclitaxel Eluting Stent With Biodegradable Polymer Versus an Uncoated Bare Metal Stent. A Prospective, Multicentric and Randomized Study.(EUCATAX Trial)
Brief Title: A Trial Comparing a Paclitaxel Eluting Stent With Biodegradable Polymer Versus a Bare Metal Stent
Acronym: EUCATAX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro de estudios en Cardiologia Intervencionista (Other)
Collaborators: Eucatech AG (Industry)
Responsible Party: Alfredo E Rodriguez, MD, PHD, FACC, FSCAI, Centro de Estudios en Cardiologia Intervencionista
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02-CECI; 02-CECI; IMA 01 (Other: Clinica IMA, Buenos Aires, Argentina)
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2010-05

CONDITIONS: Coronary Artery Disease
Keywords: Biodegradable polymer; Drug Eluting Stent; In stent restenosis; stent thrombosis; Bare Metal Stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Drug-Eluting Stents

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1-BMS (Active Comparator): Bare Metal Stent (Euca STS Flex)
  Interventions: Device: Bare Metal Stent
- 2-DES (Experimental): Drug Eluting Stent (Euca STS Flex DE), Paclitaxel Eluting stent with biodegradable polymer
  Interventions: Device: Drug Eluting Stent

INTERVENTIONS:
Device: Bare Metal Stent — Stainless steel stent
  Other Names: Euca STS Flex
  Arms: 1-BMS
Device: Drug Eluting Stent — stent coated with the biodegradable polymer matrix hemoparin and paclitaxel
  Other Names: Euca STS Flex DE
  Arms: 2-DES

SUMMARY:
The success of stent implantation has led to the increasingly widespread use of them in the treatment of coronary artery disease (Sigwart, Serruys, Fischman)and although stent restenosis is still a limit for this therapeutic mode (Serruys, Rodriguez) the new generation of stents with improved coating materials and the development of polymers that release different kinds of drugs that prevent the activation and/or proliferation of smooth muscle cells (ultimate cause of restenosis) (Grube, Rodriguez). shows major improvements on this matter. The new generation of stents with biodegradable polymers and short time of drug release gives new advantages to this therapeutic, multiple studies and registries challenge this new devices (Taxus I and II, RAVEL, SIRIUS, ERACI II and III).

For this reason the present study aims to compare a stainless steel stent with a drug eluting stent with coated of biodegradable polymer matrix hemoparin and paclitaxel.

DETAILED DESCRIPTION:
Patients with de novo lesions treated in different Institutions in Buenos Aires Argentina were randomized to treat with a stainless steel stent ("euca STS Flex") or a drug-eluting stent (" euca STS Flex DE") with a coating of a biodegradable polymer matrix of hemoparin and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Patient signing informed consent after receiving extensive written and oral information about the trial,
* Older than 18 years,
* Agreement to have a control examination done after six months,
* Patients with angina pectoris symptoms (CCS stages i-IV, unstable angina pectoris Braunwald B and C) and patients with documented silent ischemia;
* Patients with one or more de novo lesions which all are to be dilated in the same session;
* Target vessel diameter of 2.5 to 4.0 mm

Exclusion Criteria:

* Female patients of child bearing age with pregnancy suspicion(a pregnancy test will be done in this cases)
* Acute myocardial infarction (Q wave or non Q wave ) with documented CK levels more than 2 fold higher than the normal values in the preceding 72 hours ,
* Substantially calcified lesion precluding successful pre dilatation,
* Ejection Fraction less than 35%,
* Patient with previous PCI with one DES,
* Target lesion < 2.5 mm
* Coagulopathy or clotting disorders, leucopenia anemia or thrombocytopenia,
* Allergy, hypersensitivity or adverse reaction to paclitaxel,
* Intolerance to the clopidogrel, Ticlopidine or Aspirin or unable to receive clopidogrel for one year,
* Active duodenal or gastric ulcer,
* Life Expectancy less than 1 year,
* Patient with LM disease (>50%)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure | six months

SECONDARY OUTCOMES:
Stent thrombosis | one year
Paclitaxel allergy | six months
Cost-effectiveness | one year
Quantitative Coronary Angiography | six months

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo E Rodriguez, MD, PHD, Study Chair — Centro de estudios en Cardiologia Intervencionista; Carlos Fernandez-Pereira, MD, Study Director — Centro de estudios en Cardiologia Intervencionista; Alfredo E Rodriguez, MD, PHD, Principal Investigator — Centro de Estudios en Cardiologia Internvencionista
Locations (2):
- Argentina (2):
  - Clinica IMA, Adrogué, Buenos Aires
  - Sanatorio Otamendi y Miroli, Buenos Aires, Buenos Aires

REFERENCES:
- [Background] Sigwart U, Puel J, Mirkovitch V, Joffre F, Kappenberger L. Intravascular stents to prevent occlusion and restenosis after transluminal angioplasty. N Engl J Med. 1987 Mar 19;316(12):701-6. doi: 10.1056/NEJM198703193161201. PMID 2950322
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Serruys PW, Unger F, Sousa JE, Jatene A, Bonnier HJ, Schonberger JP, Buller N, Bonser R, van den Brand MJ, van Herwerden LA, Morel MA, van Hout BA; Arterial Revascularization Therapies Study Group. Comparison of coronary-artery bypass surgery and stenting for the treatment of multivessel disease. N Engl J Med. 2001 Apr 12;344(15):1117-24. doi: 10.1056/NEJM200104123441502. PMID 11297702
- [Derived] Rodriguez AE, Vigo CF, Delacasa A, Mieres J, Fernandez-Pereira C, Bernardi V, Bettinoti M, Rodriguez-Granillo AM, Rodriguez-Granillo G, Santaera O, Curotto V, Rubilar B, Tronge J, Palacios IF, Antoniucci D; EUCATAX Investigators. Efficacy and safety of a double-coated paclitaxel-eluting coronary stent: the EUCATAX trial. Catheter Cardiovasc Interv. 2011 Feb 15;77(3):335-42. doi: 10.1002/ccd.22769. Epub 2010 Nov 30. PMID 20824769
- See also: German Cardiac Society — http://www.dgk.org
- See also: Centro de Estudios en Cardiologia Intervencionista — http://www.centroceci.com.ar